CLINICAL TRIAL: NCT04281160
Title: Patient Centered Outcomes Analysis for MS Using a Mobile Application
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: BeCare Link LLC (Industry)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1608017501
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis
Keywords: mobile app; TUG test; 25 foot walk; six minute walk; working memory test; Contrast Sensitivity; Coded Message Cognitive Test; Fine motor function; Digit Modality test
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Metric: Patients and healthy controls were evaluated by expert raters with standard clinical metrics of neurologic function.
  Interventions: Device: BeCare Mobile App
- Mobile Activity Metric: Patient performed mobile activity
  Interventions: Device: BeCare Mobile App

INTERVENTIONS:
Device: BeCare Mobile App — The BeCare App is a mobile application that will perform routine assessments of neurological function in individuals with MS and address the most relevant domains that are affected in MS: cognition, afferent visual functioning, motor functioning, fine motor functioning, coordination, gait, and endurance

SUMMARY:
Multiple Sclerosis (MS) is a demyelinating disease of the central nervous system (CNS) that can impact all aspects of nervous system function. Currently clinical assessments as part of the standard of care are performed in the health care providers office during regularly scheduled visits and are semi-quantitative or qualitative in nature. The goal of the BeCare Multiple Sclerosis Assessment App is to allow for patient centered, frequent, and quantitative assessments of neurologic function through a mobile App. The BeCare MS App integrates with all Android and Apple operating systems. The investigator's overall goal is to improve well-being of people with MS through accurate assessment of their neurologic function to be used by themselves as well as their health care providers. The purpose of this Clinical Trial is to validate the App based assessments versus Gold-Standard clinical assessments.

DETAILED DESCRIPTION:
Patients will complete the 11 App based and clinically based assessments in one visit. These will be repeated 3-7 times to eliminate learning variation. The assessments and the instructions to complete these assessments are on the App and listed below.

1. Timed Up and Go (TUG). The primary endpoint of this study is to compare the App-based TUG with the clinically derived TUG results. The hypothesis is that the App based result and the clinically derived result are equivalent. The TUG is a validated assessment of functional mobility (2). For the TUG, the Subject is seated in a regular chair with no chair arm-rests. At the start of the test designated by a vocal cue, the Subject will stand walk to a mark three meters from where there feet are placed when sitting, turn 180 degrees, walk back to the chair and sit to finish. The test result is recorded as the time from start to finish. Normative data have been established for the TUG and the test has been validated in MS (2). For the App-based assessment the Subject will hold their mobile devise in their hand, they will select on the test and then perform the test without external cue. For the traditional TUG, the subject will be instructed to start by a research coordinator who will also start a timer. The research coordinator will stop the timer when the Subject has seated. During the traditional TUG test the Subject will also be holding their mobile phone in their hand as they had done for the App-based test. Three comparisons will be made: App-based result when the Subject self-initiates versus the traditional result; App-based result when the patient self initiates versus the App-based result when the patient is instructed to start; ands App-based result when the patient is instructed to start versus the traditional result. A students t-test or a Welch's t-test will be performed with a Bonferroni correction when indicated.
2. Fine motor function/rapid finger movements (FMF) is a secondary endpoints. FMF is assessed by having the patient tap the interphalangeal crease of their thumb with the ipsilateral index finger tip. This movement is typically impacted with upper motor neuron dysfunction, cerebellar dysfunction, and possibly with severe loss of position sense and is a sensitive indicator of dysfunction. However, this test is never quantitatively reported in the neurologic exam. For the traditional test, patients will be asked to tap their finger on their thumb crease as rapidly as possible for 10 seconds. The test will be reported as normal, slowed, or severely impaired. The normal variation between dominant and non-dominant hands will be noted. For the App based test the Subject will be presented with a game on their mobile phone that requires them to tap a designated spot as frequently as possible for 10 seconds. The phone will record the number of taps, the regularity of their spacing and any consistent change over time (fatigue). The test will be repeated 3 times and results presented as the mean +/- SD for each measurement. The change in frequency over time will be reported. A students t-test or a Welch's t-test will be performed with a Bonferroni correction when indicated.
3. Upper extremity coordination (secondary endpoint). Upper extremity cerebellar function is typically measured doing a finger-nose-finger test where the subject touches the examiners finger, then their own nose, then the examiners finger again. Typically, the movement is repeated several times. In the clinical setting, the test is commonly reported as normal, impaired (mild dysmetria) or severely impaired (marked dysmetria). For the App based test, the Subject will be asked to move an object with their index finger such that it stays within the boundaries of a moving path. The App will measure deviations outside the path as well as circumstances in which these deviations occur. The test will be repeated 3 times on each side and results presented as the mean for each deviation greater than 2 standard deviations in difference from the control population. The change in frequency over time will be reported as the XXXX. A students t-test or a Welch's t-test will be performed with a Bonferroni correction when indicated.
4. Auditory-Comprehension-Typing (ACT) test (secondary endpoint). In this test the subject is given a short auditory phrase and then must type that phrase using a virtual keyboard. The time to complete typing the phrase as well as the time interval and time variance between keystrokes is compiled and compared to healthy age-matched controls. To control for fine motor function the virtual keyboard records the time and variance for tapping a series of keys that spontaneously change color (white background to green for example), which is termed the maximal keystroke velocity (strokes/second). [should the maximal keystroke velocity be subtracted or used as a denominator?] Comparisons are made between Subjects and Healthy controls for the absolute time to type the phrase, and for the key-stroke variance. Harmonic and conjugate harmonic functions will be determined by the Milne - Thompson method and expressed in a two-dimensional surface.
5. Timed 25-foot walk (secondary endpoint). At the start of the test the subject is standing at a mark (typically taped on the floor) and is prepared to walk to the destination mark 25 feet away. Timing begins with a vocal cue and the Subject walks as quickly as possible while remaining safe, to the 25 foot mark. The test result is recorded as the time from start to finish. Normative data have been established for the Timed 25 foot walk and the test has been validated in MS (3). For the App-based assessment the Subject will hold their mobile devise in their hand, they will select the test and then perform the test without external cue. For the traditional Timed 25 foot walk, the subject will be instructed to start by a research coordinator who will also start a timer. The research coordinator will stop the timer when the Subject has reached the 25-foot mark. Three comparisons will be made: App-based result when the Subject self-initiates versus the traditional result; App-based result when the patient self initiates versus the App-based result when the patient is instructed to start; and the App-based result when the patient is instructed to start versus the traditional result. A students t-test or a Welch's t-test will be performed with a Bonferroni correction when indicated.
6. Coded Message Cognitive Test (secondary endpoint). For this test the subject is asked to decode a message using decoding key. A series of symbols are paired with letters or words to be used as the key. The coded message is provided in symbols. The Subject self starts the test by pressing a "begin button" and the test stops when the Subject completes the decoded message. For the standard test, subjects will perform the symbol digit modality test. Normative data for the Coded Message Cognitive test will be generated. Comparisons will be maded between MS Subjects and the normative data for the Coded Message Test, as well as between the Coded Message Test and the Symbol Digit Modality test.
7. Six minute walk (secondary endpoint). For this test we will measure the distance covered by the Subject while walking at a comfortable and safe pace for 6 minutes. The App will record distance using GPS and will record the number of steps taken using the mobile devises accelerometer. This test will be performed once with the observation of a research coordinator and then three additional times within three days time by the subject. Mean times and mean step numbers will be determined and compared to normative data.
8. Contrast Sensitivity (secondary endpoint). For this test the subject is asked to discern or read letters/numerals off a screen with varying contrast sensitivity (grey on grey). Next to each letter/number is a box for them to enter the character/numeral using a virtual keyboard. The number of correct assignments are recorded and reported as a fraction of the total number tested. For the standard test, subjects are asked to report the numbers or letters of a standard Snellen chart as well as low contrast Snellen charts (2.5, 1.25). Comparisons will be made between the subject and the normative data for each test. Comparisons will also be made between normalized values for each test for each Subject. A third test will be performed in which the subject "rolls" a ball through a maze of ever decreasing contrast sensitivity. The size of the maze path will be adjusted based on their cerebellar and fine motor function determined above. The time to first error and the time to repeated errors is determined.
9. Arm Swing Test (secondary endpoint). For this test the subject is asked to hold their mobile device in their dominant hand and then raise their arms to pass the devise to their other hand over the top of their head. This is repeated as fast as possible for 30 seconds. For the standard test, upper extremity strength is recorded on the neurologic 5 point scale (5 = normal, 4 = active resistance, 3 = antigravity, 2 = movement in the absence of gravity, 1 = movement of a muscle but no movement of the limb, 0 = no movement at all. Comparisons will be made between each subject and normative data, and between the two test groups.
10. Birds in a box working memory test (secondary). For this test the subject is presented with 5 boxes in a row, each with a different colored bird in them and told to memorize the bird color for each box. After 8 seconds, the boxes are closed and above one box five bird color choices will appear at which time the subject must place a new bird in that box without violating the rule that the original 5 boxes in a row can not have more than two birds of the same color at any one time. The appearance of birds to drop into the box will be mathematically determined to pose the same risk/difficulty for each subject. The number of errors are recorded and the number of correct choices are recorded over 90 seconds. For the standard test, subjects will perform the Paced Serial Addition Test (PASAT). PASAT and Birds in a box results will be normalized and compared for each subject. If the subject has difficulty with fine motor function, a normalization factor will be provided to increase the time to complete the task.
11. Balance Test (secondary). The subject is asked to stand with feet together and then raise their non-dominant leg such that their knee is at waist level. The time is recorded until the patient looses balance and touches the ground with the raised foot. The test is repeated for a total of three times for each side alternating for side to side. Test results are compared to healthy controls to achieve normative data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with multiple sclerosis- male and female patients between the ages of 18 and 65 who have been accurately diagnosed with MS based on the revised MacDonald criteria
2. Subjects must have the ability to provide consent and be willing to participate in the study.
3. Participants- both MS subjects and healthy subjects- must self-report having a smartphone on which they can download the BeCare application

Exclusion Criteria:

1. Subjects must not have a history of concurrent illnesses that result in physical or cognitive disability such as rheumatoid arthritis, osteoarthritis, and Alzheimer's Disease.
2. Chronic, clinically significant (unresolved, requiring on-going medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality, self reported
3. Subjects who do not own a smartphone in which they can download the BeCare application will be excluded from this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 60 participants will take part in this study: 40 participants with mild to moderate MS and 20 participants without MS will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Compare the App-based TUG with the clinically derived TUG results | 6 months
  The Subject is seated in a regular chair with no chair arm-rests. The Subject will stand and then walk to a mark three meters away, turn 180 degrees, walk back to the chair and sit to finish. The test result is recorded as the time from start to finish. For the App-based assessment the Subject will hold their mobile devise in their hand, select the TUG test and then perform the test without external cue. For the traditional TUG, the subject will be instructed to start by a research coordinator who will also start a timer. The research coordinator will stop the timer when the Subject has seated. Three comparisons will be made: App-based result when the Subject self-initiates versus the traditional result; App-based result when the patient self initiates versus the App-based result when the patient is instructed to start; ands App-based result when the patient is instructed to start versus the traditional result.

SECONDARY OUTCOMES:
Fine motor function/rapid finger movements (FMF) | 6 months
  FMF is assessed by having the patient tap the interphalangeal crease of their thumb with the ipsilateral index finger tip. This movement is typically impacted with upper motor neuron dysfunction, cerebellar dysfunction, and possibly with severe loss of position sense and is a sensitive indicator of dysfunction. For the traditional test, patients will be asked to tap their finger on their thumb crease as rapidly as possible for 10 seconds. The normal variation between dominant and non-dominant hands will be noted. For the App based test the Subject will be presented with a game on their mobile phone that requires them to tap a designated spot as frequently as possible for 10 seconds. The phone will record the number of taps, the regularity of their spacing and any consistent change over time (fatigue). The test will be repeated 3 times and results presented as the mean +/- SD for each measurement. The change in frequency over time will be reported.
Upper extremity coordination | 6 months
  Upper extremity cerebellar function is typically measured doing a finger-nose-finger test where the subject touches the examiners finger, then their own nose, then the examiners finger again. Typically, the movement is repeated several times. In the clinical setting, the test is commonly reported as normal, impaired (mild dysmetria) or severely impaired (marked dysmetria). For the App based test, the Subject will be asked to move an object with their index finger such that it stays within the boundaries of a moving path. The App will measure deviations outside the path as well as circumstances in which these deviations occur. The test will be repeated 3 times on each side and results presented as the mean for each deviation greater than 2 standard deviations in difference from the control population. The change in frequency over time will be reported.
Auditory-Comprehension-Typing (ACT) test | 6 months
  The subject is given a short auditory phrase and then must type that phrase using a virtual keyboard. The time to complete typing the phrase as well as the time interval and time variance between keystrokes is compiled and compared to healthy age-matched controls. To control for fine motor function the virtual keyboard records the time and variance for tapping a series of keys that spontaneously change color (white background to green for example), which is termed the maximal keystroke velocity (strokes/second). [should the maximal keystroke velocity be subtracted or used as a denominator?] Comparisons are made between Subjects and Healthy controls for the absolute time to type the phrase, and for the key-stroke variance. Harmonic and conjugate harmonic functions will be determined by the Milne - Thompson method and expressed in a two-dimensional surface.
Timed 25-foot walk | 6 months
  The subject is standing at a mark (taped on the floor) and is prepared to walk to the destination mark 25 feet away. Timing begins with a vocal cue and the Subject walks as quickly as possible while remaining safe, to the 25 foot mark. The test result is recorded as the time from start to finish. For the App-based assessment the Subject will hold their mobile devise in their hand, they will select the test and then perform the test without external cue. For the traditional Timed 25 foot walk, the subject will be instructed to start by a research coordinator who will also start a timer, and will stop the timer when the Subject has reached the 25-foot mark. Three comparisons will be made: App-based result when the Subject self-initiates versus the traditional result; App-based result when the patient self initiates versus the App-based result when the patient is instructed to start; and the App-based result when the patient is instructed to start versus the traditional result.
Coded Message Cognitive Test | 6 months
  The subject is asked to decode a message using decoding key. A series of symbols are paired with letters or words to be used as the key. The coded message is provided in symbols. The Subject self starts the test by pressing a "begin button" and the test stops when the Subject completes the decoded message. For the standard test, subjects will perform the symbol digit modality test. Normative data for the Coded Message Cognitive test will be generated. Comparisons will be made between MS Subjects and the normative data for the Coded Message Test, as well as between the Coded Message Test and the Symbol Digit Modality test.
Six minute walk | 6 months
  we will measure the distance covered by the Subject while walking at a comfortable and safe pace for 6 minutes. The App will record distance using GPS and will record the number of steps taken using the mobile devises accelerometer. This test will be performed once with the observation of a research coordinator and then three additional times within three days time by the subject.
Contrast Sensitivity | 6 months
  The subject is asked to discern or read letters/numerals off a screen with varying contrast sensitivity (grey on grey). Next to each letter/number is a box for them to enter the character/numeral using a virtual keyboard. The number of correct assignments are recorded and reported as a fraction of the total number tested. For the standard test, subjects are asked to report the numbers or letters of a standard Snellen chart as well as low contrast Snellen charts (2.5, 1.25). Comparisons will be made between the subject and the normative data for each test. Comparisons will also be made between normalized values for each test for each Subject. A third test will be performed in which the subject "rolls" a ball through a maze of ever decreasing contrast sensitivity. The size of the maze path will be adjusted based on their cerebellar and fine motor function determined above. The time to first error and the time to repeated errors is determined
Arm Swing Test | 6 months
  The subject is asked to hold their mobile device in their dominant hand and then raise their arms to pass the devise to their other hand over the top of their head. This is repeated as fast as possible for 30 seconds. For the standard test, upper extremity strength is recorded on the neurologic 5 point scale (5 = normal, 4 = active resistance, 3 = antigravity, 2 = movement in the absence of gravity, 1 = movement of a muscle but no movement of the limb, 0 = no movement at all. Comparisons will be made between each subject and normative data, and between the two test groups.
Birds in a box working memory test | 6 months
  For this test the subject is presented with 5 boxes in a row, each with a different colored bird in them and told to memorize the bird color for each box. After 8 seconds, the boxes are closed and above one box five bird color choices will appear at which time the subject must place a new bird in that box without violating the rule that the original 5 boxes in a row can not have more than two birds of the same color at any one time. The appearance of birds to drop into the box will be mathematically determined to pose the same risk/difficulty for each subject. The number of errors are recorded and the number of correct choices are recorded over 90 seconds. For the standard test, subjects will perform the Paced Serial Addition Test (PASAT). PASAT and Birds in a box results will be normalized and compared for each subject. If the subject has difficulty with fine motor function, a normalization factor will be provided to increase the time to complete the task.

CONTACTS AND LOCATIONS:
Overall Officials: Larry D Rubin, MPh, Study Director — Sponsor GmbH
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berrigan LI, Fisk JD, Walker LA, Wojtowicz M, Rees LM, Freedman MS, Marrie RA. Reliability of regression-based normative data for the oral symbol digit modalities test: an evaluation of demographic influences, construct validity, and impairment classification rates in multiple sclerosis samples. Clin Neuropsychol. 2014;28(2):281-99. doi: 10.1080/13854046.2013.871337. Epub 2014 Jan 20. PMID 24438521
- [Result] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Result] Sebastiao E, Sandroff BM, Learmonth YC, Motl RW. Validity of the Timed Up and Go Test as a Measure of Functional Mobility in Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2016 Jul;97(7):1072-7. doi: 10.1016/j.apmr.2015.12.031. Epub 2016 Mar 2. PMID 26944709